CLINICAL TRIAL: NCT01782443
Title: Phase II Study of Ziv-aflibercept in Patients With Advanced, Progressive Carcinoid Tumors
Brief Title: Ziv-Aflibercept for Advanced Progressive Carcinoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Chan, MD, MPH, Prinicipal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-456
Record Dates: First submitted 2013-01-31; First posted 2013-02-01 (Estimated); Results first posted 2022-11-09 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Carcinoid Tumor
Keywords: Progressive; Metastatic
MeSH Terms: conditions — Carcinoid Tumor; Neoplasm Metastasis | interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental Treatment Arm (Experimental): Ziv-aflibercept IV every 2 weeks, 4 mg/kg
  Interventions: Drug: Ziv-aflibercept

INTERVENTIONS:
Drug: Ziv-aflibercept

SUMMARY:
This research study is a Phase II clinical trial, which tests the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific cancer. "Investigational" means that the drug, Ziv-aflibercept, is being studied. It also means that the FDA has not yet approved Ziv-aflibercept for use in patients with your type of cancer.

Every person has molecules in their bloodstream called vascular endothelial growth factors (VEGFs). These molecules help grow and sustain new blood vessels needed by the human body. Cancer tumors hijack this mechanism because they need new blod vessels and oxygen to grow. Ziv-aflibercept is an antibody. Antibodies are proteins that are produced naturally in our bodies and help to recognize foreign substances in our body. Ziv-aflibercept is a "targeted therapy" called a "VEGF Trap", that "traps" (binds) these VEGFs and prevents the cancer from using them to grow.

Though Ziv-aflibercept has not yet been FDA approved for the treatment of carcinoid tumors, it has recently been approved for patients with treatment-resistant colorectal cancer.

In this research study, we will use Ziv-aflibercept in combination with standard octreotide therapy to see if it slows the growth or spread of your carcinoid tumor. Standard octreotide (sandostatin) therapy is currently approved for treating symptoms of carcinoid tumors, such as those caused by carcinoid syndrome. Carcinoid syndrome is caused by hormones and other substances released by carcinoid tumors into the bloodstream. One of these secreted substances is serotonin, one of the body's natural chemical messengers. When excess serotonin secreted by the carcinoid tumors reaches the body's tissues, it is thought to cause diarrhea and redness (flushing) of the face, chest or back. Excess serotonin may also cause changes in the structure of the heart valves, which can impair the heart's function. Octreotide works by binding to receptors found on carcinoid tumors and prevents the release of hormones from the tumor.

DETAILED DESCRIPTION:
If you are willing to participate in this study you will be asked to undergo some screening tests and procedures to confirm that you are eligible. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that you do not take part in the research study. If you have had some of these tests or procedures recently, they may or may not have to be repeated. These tests and procedures include: a medical history, physical examination, CT or MRI, blood tests, serum chromogranin A, urine tests, 24-hour urine collection, pregnancy test and an electrocardiogram. If these tests show that you are eligible to participate in the research study, you will begin the study treatment. If you do not meet the eligibility criteria, you will not be able to participate in this research study.

If you meet the requirements for this study and you agree to continue your participation, you will receive Ziv-aflibercept every two weeks. Each dose of Ziv-aflibercept consists of an approximately 60 minutes infusion (through a needle into a vein). You will also receive an injection of Octreotide LAR (long acting release) monthly as part of your treatment for carcinoid tumor. This injection will be given to you by a nurse in your buttock. You may already be on Octreotide LAR. In that case, you will continue taking it at the same dose and schedule.

You will need to come to the clinic every two weeks while participating in this study. Each cycle is 28 days.

The following tests and procedures will be performed on Days 1 and 15 of each cycle: questions about your health, physical exam (Day 1 of each cycle only), vital signs, blood tests, pregnancy test (Day 1 of each cycle only).

Urine tests will be performed every other cycle.

The following tests and procedures will be done at the end of every third cycle: CT scan or MRI, Serum Chromogranin A, 24-hour urine collection.

After the final dose of the study drug the following tests and procedures will be performed: questions about your general health, physical exam, vital signs, blood tests, pregnancy test, EKG, Serum Chromogranin A, 24-hour urine collection.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed well differentiated or moderately differentiated neuroendocrine tumor from either a primary or metastatic site
* Must have disease that is not amenable to curative resection
* Must have evidence of disease progression within 12 months prior to study entry
* Must have measurable disease (RECIST 1.1)
* Prior chemoembolization of local ablative therapies are allowed, provided there is measurable disease outside of the area treated, or documented evidence of progression at the site of prior treatment
* No limit to number of prior treatments. Prior bevacizumab allowed unless discontinued due to unacceptable toxicity. Prior TKI targeting VEGF receptors allowed
* Treatment with a somatostatin analog required for all subjects
* Subjects with history of hypertension must be adequately controlled
* Therapeutic anticoagulation is allowed. Must be on a stable dose of anticoagulant medication
* Must agree to use adequate contraception prior to study entry, for the duration of study participation and for 3 months after last administration of study drug

Exclusion Criteria:

* Prior treatment including chemoembolization within 4 weeks of study entry
* Major surgery within 4 weeks of study entry or minor surgery within 2 weeks of study entry
* Pregnant or breastfeeding
* Poorly differentiated carcinoma, high grade neuroendocrine tumor or small cell carcinoma
* Prior treatment with Ziv-aflibercept
* Pancreatic neuroendocrine tumor (islet cell carcinoma)will be excluded from this study. All non functional and functional islet cell carcinomas such as insulinoma, glucagonoma, gastrinoma, VIPoma will be excluded.
* Not adequately recovered from toxicity of previous therapy
* Known untreated brain or other central nervous system metastases
* Known allergy to any of the study agents or to compounds of similar chemical or biologic composition
* History of congestive heart failure
* Symptomatic peripheral arterial disease
* Unhealed wounds, ulcers or bone fractures
* HIV positive or active Hepatitis infection
* History of abdominal fistula, GI perforation, intra abdominal abscess, uncontrolled GI bleeding, diverticulitis within 6 months of study entry
* History of arterial thrombotic events such as myocardial infarction, unstable angina pectoris or any ischemic or hemorrhagic cerebrovascular accident within the past 6 months
* No history of pulmonary embolism, DVT or vascular access related thrombosis if not also receiving adequate anticoagulation at a stable dose.
* No history of prior or synchronous malignancy except if treated with curative intent at least 3 years prior to study entry, or adequately treated non-melanoma skin cancer, cervical carcinoma in situ, or prostate intraepithelial neoplasia without evidence of prostate cancer
* Uncontrolled non-malignant illness that may increase the risks associated with study participation or may interfere with the conduct of the study or interpretation of study results
* Uncontrolled psychiatric illness or social situations that would limit compliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-02-13 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Chan, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Perez K, Kulke MH, Horick NK, Regan E, Graham C, Scheutz S, Stonely D, Enzinger PC, Fuchs CS, Allen JN, Enzinger AC, Clark JW, Chan JA. A Phase II Study of Ziv-Aflibercept in Patients With Advanced Extrapancreatic Neuroendocrine Tumors. Pancreas. 2022 Aug 1;51(7):763-768. doi: 10.1097/MPA.0000000000002099. PMID 36395401

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental Treatment Arm (Ziv-aflibercept): Ziv-aflibercept IV every 2 weeks, 4 mg/kg for the first 10 patients, 2 mg/kg for the remaining 9 patients
Period: Overall Study
Arm/Group | Experimental Treatment Arm (Ziv-aflibercept)
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental Treatment Arm (Ziv-aflibercept)
Number analyzed (Participants) | 19
Age, Continuous [Median (Full Range); unit: years] | 61 [48 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 19
primary site [Count of Participants; unit: Participants]
  midgut | 12
  unknown | 4
  rectum | 1
  lung | 1
  thymus | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: To evaluate the progression-free survival (PFS) duration of patients with metastatic, unresectable, progressive carcinoid tumors treated with Ziv-aflibercept. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) was used.
  Progressive Disease (PD) is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study with at least a 5 mm absolute increase in the sum of all lesions. The appearance of one or more new lesions denotes disease progression. Partial Response (PR) is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: 2 years
Population: The efficacy of ziv-aflibercept was evaluated amongst all patients who were treated on protocol (4 mg/kg in 10 patients, reduced to 2 mg/kg in 9 patients due to adverse events observed at the higher does level).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental Treatment Arm (Ziv-aflibercept)
Number analyzed (Participants) | 19
months | 11.8 [3.2 to 16.1]

2. Secondary Outcome: Evaluation of Disease Response
Description: To evaluate disease response using RECIST criteria, version 1.1, of patients with advanced carcinoid tumors treated with Ziv-aflibercept.
  Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI or CT include the following categories of disease response: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable disease (SD), less than 30% decrease but no more than 20% increase in sum of the longest diameter of target lesions.
Time Frame: 2 years
Population: 14 patients were evaluated for disease response per RECIST 1.1. The remaining 5 patients were not evaluable for response by RECIST 1.1 because they did not undergo protocol restaging due to early withdrawal from the study prior to reaching first protocol restaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Arm (Ziv-aflibercept)
Number analyzed (Participants) | 14
Participants
  Partial Response | 1
  Stable Disease | 13

3. Secondary Outcome: Evaluation of Biochemical Response - Number of Patients With Greater Than 50% Drop in Chromogranin A From Baseline
Description: To evaluate biochemical response in patients with elevated chromogranin A at baseline, using levels of chromogranin-A measured at baseline and following treatment with Ziv-aflibercept. Biochemical response was defined as greater than 50% drop in chromogranin A from baseline.
  During the screening period, all patients were evaluated for serum chromogranin A. Per protocol, if results of these are normal at baseline, they were not repeated while on study. If above institutional ULN at baseline, they were evaluated at time of tumor restaging.
Time Frame: 2 years
Population: 12 participants were evaluable based on baseline assessment of serum chromogranin A. These patients were evaluated for a greater than 50% drop in chromogranin A from baseline while on treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Arm (Ziv-aflibercept)
Number analyzed (Participants) | 12
Participants | 2

4. Secondary Outcome: Biochemical Response - Number of Patients With Greater Than 50% Drop in 24hr Urine 5-HIAA From Baseline
Description: To evaluate biochemical response in patients with elevated 24hr urine 5-HIAA at baseline, using levels of 24hr urine 5-HIAA at baseline and following treatment with Ziv-aflibercept. Biochemical response was defined as greater than 50% drop in 24hr urine 5-HIAA from baseline.
  During the screening period, all patients were evaluated for 24hr urine 5HIAA. Per protocol, if results of these were normal at baseline, they were not repeated while on study. If above institutional ULN at baseline, they were evaluated at time of tumor restaging.
Time Frame: 2 years
Population: 11 patients were evaluable based on baseline assessment of 24hr urine 5-HIAA. These patients were followed for greater than 50% drop in 24hr urine 5-HIAA after starting treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Treatment Arm (Ziv-aflibercept)
Number analyzed (Participants) | 11
Participants | 1

ADVERSE EVENTS:
Time Frame: Patients were followed for AEs from first dose of study treatment, throughout the study, and through 30 days of the last study treatment, an average of 16 months. Participants removed from study for unacceptable adverse events were followed until resolution or stabilization of the adverse event.
Description: Adverse Event (AE): An adverse event (AE) is any untoward medical occurrence in a patient administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. Abnormal laboratory values or diagnostic test results constitute adverse events only if they are determined to be of clinical significance or require treatment or further diagnostic tests. Adverse events are reported for all patients, based on starting dose
Groups:
- Ziv-aflibercept 4mg/kg: Patients treated with a starting dose of Ziv-aflibercept 4 mg/kg
- Ziv-aflibercept 2mg/kg: Patients treated with a starting dose of Ziv-aflibercept 2 mg/kg
Arm/Group | Ziv-aflibercept 4mg/kg | Ziv-aflibercept 2mg/kg
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/10 | 5/9
Other Adverse Events (participants affected / at risk) | 10/10 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ziv-aflibercept 4mg/kg (N=10) | Ziv-aflibercept 2mg/kg (N=9)
Hypertension (Cardiac disorders) | 2 | 1
Reversible Cerebral Vasoconstriction Syndrome (Nervous system disorders) | 1 | 0
Mouth sores (Gastrointestinal disorders) | 1 | 0
pain (General disorders) | 0 | 3
pneumonia (Infections and infestations) | 0 | 1
death due to disease progression (General disorders) | 1 | 0
Intracranial bleeding (Nervous system disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ziv-aflibercept 4mg/kg (N=10) | Ziv-aflibercept 2mg/kg (N=9)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Anorexia (General disorders) | 2 | 2
diarrhea (Gastrointestinal disorders) | 1 | 1
fatigue (General disorders) | 5 | 3
hypertension (Cardiac disorders) | 9 | 9
headache (Nervous system disorders) | 1 | 2
subarachnoid hemorrhage (Nervous system disorders) | 1 | 0
stroke (Nervous system disorders) | 1 | 0
palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 | 1
proteinuria (Renal and urinary disorders) | 1 | 3
alkaline phosphatase increased (Gastrointestinal disorders) | 0 | 1
creatinine increase (Renal and urinary disorders) | 0 | 1
hoarseness (General disorders) | 0 | 2
confusion (Nervous system disorders) | 0 | 1
flushing (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-21): https://cdn.clinicaltrials.gov/large-docs/43/NCT01782443/Prot_SAP_000.pdf